CLINICAL TRIAL: NCT03655314
Title: Beginning With a Healthy Start: A Randomized Controlled Trial of Informatics-Enhanced Newborn Weight Management
Brief Title: Using the Electronic Health Record to Guide Management of Newborn Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-23249
Record Dates: First submitted 2018-08-27; First posted 2018-08-31 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive; Morbidity;Perinatal; Feeding, Bottle
Keywords: formula
MeSH Terms: conditions — Breast Feeding; Bottle Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newborn Weight Tool (NEWT) (Active Comparator): The electronic medical record will display the Newborn Weight Tool along with a banner flagging newborn weight loss greater than or equal to the 75th centile of birth weight
  Interventions: Other: NEWT
- Usual care (Placebo Comparator): As with usual care, the electronic medical record will display the weight only as weight in grams and percent weight lost from birth weight
  Interventions: Other: Usual care

INTERVENTIONS:
Other: NEWT — The Newborn Weight Tool (NEWT) is publicly available at www.newbornweight.org. For this intervention, NEWT will be embedded into the electronic medical record along with a flag for weight loss greater than or equal to the 75th centile of birth weight.
  Other Names: Newborn Weight Tool
  Arms: Newborn Weight Tool (NEWT)
Other: Usual care — The electronic medical record will display the weight only as weight in grams and percent weight lost from birth weight.
  Arms: Usual care

SUMMARY:
Weight loss is normal for healthy newborns in the first few days, especially for those exclusively breastfed, who may have low enteral intake for several days. Although most newborns tolerate this early period of weight loss well, those with pronounced weight loss become at increased risk of feeding problems and hyperbilirubinemia, which are the two most common causes of neonatal readmission. To facilitate the assessment of risk for an individual newborn, the Newborn Weight Tool (NEWT) has been developed to categorize each infant's weight loss according to population norms, so that formula can be administered when weight loss is pronounced and avoided when weight loss is normal. The Healthy Start study will be a randomized, controlled trial testing whether displaying NEWT to clinicians providing newborn care can improve neonatal health outcomes including formula use, weight loss and readmission. Newborns will be randomly assigned either to display weight with NEWT weight categorization to their providers in the electronic health record (EHR) or to usual care (weight displayed without NEWT categorization).

ELIGIBILITY:
Inclusion Criteria:

* Assignment to a bed assignment on the well newborn service at the time of the first weight measured subsequent to birth weight and at >6 hours and <=96 hours of age

Exclusion Criteria:

* None

Ages: 6 Hours to 96 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2682 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Concordance with feeding recommendation during the birth hospitalization | 0-96 hours
  Feeding is defined as concordant with feeding recommendation if any of the following occur: 1) for newborns who do not have documented weight loss >=75th NEWT centile, formula is not used; 2) for newborns with only one weight documented that is more pronounced than the 75th centile, no formula is used prior to the weight documented at more pronounced than the 75th centile; 3) for newborns who have two weights documented more pronounced than the 75th centile, formula is used.

SECONDARY OUTCOMES:
Proportion readmitted to the hospital | 0-30 days
  Readmission to the hospital after discharge from the birth hospitalization
Length of hospital stay | 0-96 hours
  Length of stay during the birth hospitalization
Proportion exclusively breastfed | 0-96 hours
  Feeding only breast milk without any other fluid or food other than vitamins, minerals and medications
Proportion with donor milk use | 0-96 hours
  Use of banked donor milk
Excess neonatal outpatient utilization | 0-30 days
  >3 outpatient visits in the first 30 days (newborns may have up to 3 preventive outpatient visits in the first 30 days)
Ratio of indicated formula use to non-indicated formula use during the birth hospitalization | 0-30 days
  Ratio of formula used either for hypoglycemia or for weight loss >=75th centile to formula used for in the absence of these
Non-preventive outpatient utilization | 0-30 days
  Number of non-preventive outpatient visits
Outpatient utilization | 0-30 days
  Number of outpatient visits

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Flaherman, MD, MPH, Principal Investigator — Associate Professor of Pediatrics and Epidemiology and Biostatistics
Locations (1):
- University of California, San Francisco Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Flaherman VJ, Robinson A, Creasman J, McCulloch CE, Paul IM, Pletcher MJ. Clinical Decision Support for Newborn Weight Loss: A Randomized Controlled Trial. Hosp Pediatr. 2022 Jun 1;12(6):e180-e184. doi: 10.1542/hpeds.2021-006470. PMID 35611641